CLINICAL TRIAL: NCT01788397
Title: Effect of Comprehensive Rehabilitation at Beitostølen Healthsports Centre. A Randomized Study.
Brief Title: Effect of Comprehensive Rehabilitation at Beitostølen Healthsports Centre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beitostølen Health Sports Center (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Hakon Dalen, MD, Beitostølen Health Sports Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BHSS
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Physically Disabled
Keywords: physical disabilities; rehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity (Experimental): Physical activity 2-4 times pr. day
  Interventions: Behavioral: Physical activity
- Control group (No Intervention): No intervention in the control group

INTERVENTIONS:
Behavioral: Physical activity — Swimming, physiotherapy, water therapy, alpine skiing, xc-skiing, hippotherapy, climbing, cycling, rowing
  Other Names: Exercise
  Arms: Physical activity

SUMMARY:
The main hypothesis:

The participants receive treatment at Beitostølen within 8 weeks or within 16 weeks. The groups waiting for rehabilitation is compared with the group receiving rehabilitation

DETAILED DESCRIPTION:
nn

ELIGIBILITY:
Inclusion Criteria:

* Patients with physical disabilities admitted to treatment at BHC

Exclusion Criteria:

* Patients with severe cognitive disorders

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Quality of life | Eight weeks
  Short Form 12 v2

SECONDARY OUTCOMES:
Pain | 8 weeks
  VAS Pain
Behavioural Regulation in Exercise Questionnaire (BREQ 2) | 8 weeks
  Measures motivational regulation
Physical Activity Scale for Individuals with Physical Disabilities (PASIPD) | 8 weeks
  Measures Physical Activity level

OTHER OUTCOMES:
Self efficacy | 8 weeks
  Self-Efficacy for Managing Chronic Disease 6-Item Scale; Exercise Regularly Scale (3-item scale); Social/Recreational Activities Scale (2-item scale); Stanford Patient Education Research Centre: Lorig K, Stewart A, Ritter P, González V, Laurent D, & Lynch J, Outcome Measures for Health Education and other Health Care Interventions. Thousand Oaks CA: Sage Publications, 1996, pp.24-25,41-45.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Stalenget, Study Director — Beitostolen Healthsports Centre
Locations (1):
- Beitostolen Healtsports Centre, Beitostølen, Oppland, Norway